CLINICAL TRIAL: NCT01559350
Title: Graft Patency of the Right Coronary Artery System in OPCAB: Saphenous Vein Graft Versus Right Gastroepiploic Artery
Brief Title: Graft Patency Analysis of the Right Coronary Artery System
Status: Terminated | Type: Observational
Why Stopped: Poor recruiting rate
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-11-065
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2012-03

CONDITIONS: Coronary Artery Disease
Keywords: OPCAB
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RGEA group: A right gastroepiploic artery in situ grafting in the right coronary artery system during OPCAB
  Interventions: Procedure: A right gastroepiploic artery in situ grafting
- SVG group: A saphenous vein grafting in the right coronary artery system during OPCAB
  Interventions: Procedure: A saphenous vein grafting

INTERVENTIONS:
Procedure: A right gastroepiploic artery in situ grafting — A right gastroepiploic artery in situ grafting in the right coronary artery system during OPCAB
  Groups: RGEA group
Procedure: A saphenous vein grafting — A saphenous vein grafting in the right coronary artery system during OPCAB
  Groups: SVG group

SUMMARY:
The ideal grafts for the right coronary artery system in coronary artery bypass surgery remain controversial. The objective of this study is to compare the long-term patency of a right gastroepiploic artery and a saphenous vein graft used for revascularization of the right coronary artery system in off pump coronary artery bypass surgery and to analyze the long-term clinical outcomes.

Total 224 patients will be enrolled according to the randomization protocol.

Check list

1. Laboratories
2. Quantitative coronary analysis (preoperative)
3. Major adverse cardiac and cerebrovascular event
4. coronary CT (coronary angiography if needed) at discharge, 1, 5, 10 years postoperatively
5. Echocardiogram

5. Cardiac enzyme

DETAILED DESCRIPTION:
The ideal bypass conduit for the right coronary artery remains a subject of intense controversy. A variety of grafts and configurations are used: the right gastroepiploic artery,the right internal thoracic artery in situ or in a Y-graft configuration,the free radial artery implanted into the aorta or the left internal thoracic artery, and the saphenous vein graft. The influence of the type of graft to the right coronary artery system on clinical results remains poorly documented, and the complementary conduit of choice to this system has yet to be determined. No superior long-term patency rate for any of these grafts to the RCA has been clearly established. We have used a saphenous vein and a right gastroepiploic artery for the right coronary artery system.

ELIGIBILITY:
Inclusion Criteria:

* Angiographic evidence of severe coronary stenosis on the right coronary territory
* Elective surgery
* Isolated off pump CABG
* Age < 75 years and life expectancy > 5 years
* Preoperative RGEA diameter > 1.5mm
* Normal left ventricular function

Exclusion Criteria:

* History of upper abdomen surgery
* History of upper GI bleeding
* Active gastric or duodenal ulcer
* Body mass index > 35kg/m2
* Redo surgery
* Presence of varicose vein
* Contraindication for CABG such as malignancy or liver cirrhosis
* Other configuration than RGEA to RCA territory or SVG to RCA territory

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo OPCAB for triple vessel disease at Samsung Medical Center are enrolled.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
All cause mortality | one year

SECONDARY OUTCOMES:
Graft occlusion | one year
  Coronary CT follow up at discharge, 1, 5 and 10 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Young Tak Lee, MD, PhD, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea